CLINICAL TRIAL: NCT03685305
Title: Weight Loss and Cognitive Function in Middle-Aged and Older Adults
Brief Title: Weight Loss and Cognitive Function in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Responsible Party: Principal Investigator, Brenda Davy, Professor, Virginia Polytechnic Institute and State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18-462
Record Dates: First submitted 2018-08-27; First posted 2018-09-26 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Overweight and Obesity
Keywords: Weight loss; Cognitive function; Weight maintenance
MeSH Terms: conditions — Overweight; Obesity; Weight Loss

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypocaloric diet with hunger reduction strategy (Experimental): Participants will be prescribed a hypocaloric diet with additional instructions to promote hunger reduction. The hypocaloric diet will range 1200-1500 kcal/d, and will be based upon the 2015 US Dietary Guidelines for Americans. Dietary instructions will be provided by a Registered Dietitian.
  Interventions: Behavioral: Hypocaloric diet with hunger reduction strategy
- Hypocaloric diet without hunger reduction strategy (Active Comparator): Participants will only be prescribed a hypocaloric diet. The hypocaloric diet will range 1200-1500 kcal/d, and will be based upon the 2015 US Dietary Guidelines for Americans. Dietary instructions will be provided by a Registered Dietitian.
  Interventions: Behavioral: Hypocaloric diet without hunger reduction strategy

INTERVENTIONS:
Behavioral: Hypocaloric diet with hunger reduction strategy — Participants will be counseled to consume a hypocaloric diet during the 4-week weight loss phase. Counseling will include specific instructions on a dietary manipulation which may reduce hunger, in order to facilitate dietary adherence.This will include tracking of the strategy. They will also be provided a pedometer and instructed to attain 10,000 steps per day.
  Arms: Hypocaloric diet with hunger reduction strategy
Behavioral: Hypocaloric diet without hunger reduction strategy — Participants will be counseled to consume a hypocaloric diet during the 4-week weight loss phase. They will also be provided a pedometer and instructed to attain 10,000 steps per day.
  Arms: Hypocaloric diet without hunger reduction strategy

SUMMARY:
More than two-thirds of middle-aged and older adults are overweight, which places them at greater risk of disability and higher medical expenses. Lifestyle interventions which promote weight loss for this population are needed. However, it is not known how different weight loss approaches impact brain (cognitive) functions, such as memory and attention. The investigator's investigation aims to improve adherence to a hypocaloric diet prescription through improved attention and inhibitory control, reduced hunger, and increased satiety.

The objectives of this pilot study are to: 1) determine the feasibility and establish proof-of-concept; 2) establish proficiency and feasibility of the proposed cognitive function assessments; and 3) obtain preliminary data for effect size generation.

ELIGIBILITY:
Inclusion Criteria:

* Overweight or obese, BMI 25-40 kg/m^2
* Able to use a computer, keyboard, and mouse

Exclusion Criteria:

* Uncontrolled hypertension
* Orthopedic injury
* Other conditions that preclude participation in a walking program
* Previous participation in psychology research which involved computerized cognitive testing
* Diabetes which requires insulin

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2018-08-06 (Actual); Primary Completion 2019-08-14 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Cognitive function changes - attention | 30-min measurement per session
  Computerized tasks will score each participant's performance for attention at baseline and after both the 4-week weight loss and weight maintenance phases.
Cognitive function changes - inhibitory control | 30-min measurement per session
  Computerized tasks will score each participant's performance for inhibitory control at baseline and after both the 4-week weight loss and weight maintenance phases.
Weight change | 5-min measurement per session
  Weight will be measured on a scale at baseline and after both the 4-week weight loss and weight maintenance phases.

SECONDARY OUTCOMES:
Perceived hunger | 15-minute measurement per session
  The Visual Analog Scale (VAS) survey will be used to measure hunger at baseline and after both the 4-week weight loss and weight maintenance phases. Participants make a mark on a 100 mm line that corresponds to their subjective feelings (range of score is 0-100). The line is anchored by descriptors that are polar opposites (not at all hungry to extremely hungry). The score is determined by using the place on the line where the mark is made by the participants.

CONTACTS AND LOCATIONS:
Overall Officials: Brenda Davy, PhD, Principal Investigator — Virginia Polytechnic Institute and State University
Locations (1):
- Virginia Tech, Blacksburg, Virginia, United States